CLINICAL TRIAL: NCT07099079
Title: Post-Market Clinical Follow-up Trial to Investigate the Rotational Stability of the Hydrophobic Intraocular Lens RAO800S
Brief Title: Post-Market Clinical Follow-Up Study on the Rotational Stability of an Intraocular Lens After Cataract Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Rayner Intraocular Lenses Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: HRSS-2025-01
Record Dates: First submitted 2025-07-15; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: IOL, Cataract
MeSH Terms: conditions — Intraocular Lymphoma; Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cataract patients: Adult patients scheduled for routine bilateral cataract surgery as part of their standard clinical care. All participants receive the RayOne RAO800S non-toric monofocal intraocular lens with orientation marks.

SUMMARY:
The goal of this post-market, prospective study at multiple clinics is to evaluate the rotational stability of the RayOne Model RAO800S non-toric monofocal intraocular lens with orientation marks in adult patients undergoing cataract surgery in both eyes. The main question it aims to answer is how stable the RayOne RAO800S lens is approximately 5 months (120 to 150 days) after surgery day. Participants are adults already scheduled to undergo cataract surgery as part of clinical routine. They will be asked to attend regular follow-up visits at the clinic, where eye images will be taken to assess the rotational stability of the implanted lens.

DETAILED DESCRIPTION:
This post-market clinical follow-up (PMCF) study is a prospective, multicenter investigation in European sites. It evaluates the rotational stability of the RayOne Model RAO800S, a non-toric monofocal intraocular lens with orientation marks, following bilateral implantation. Participants will be assessed approximately 5 months (120 to 150 days) post-operatively.

ELIGIBILITY:
Eligible subjects must meet all the following inclusion criteria in both eyes.

1. Male or female, 22 years or older at the pre-operative visit who have cataract in both eyes and who are eligible for phacoemulsification cataract surgery
2. Subjects who are projected to have best corrected distance visual acuity 0.20 logMAR (20/30) or better in both eyes after IOL implantation by investigator estimation
3. Clear intraocular media other than cataract
4. Contact lens wearers must demonstrate stability of biometry in both eyes
5. Have the capability to understand and sign an EC approved informed consent form and privacy authorization in accordance with local regulations
6. Female subjects must be 1-year postmenopausal, surgically sterilized, or if childbearing potential must use a stabilized and acceptable form of contraception from the beginning throughout the end of the study.

   Stabilized and acceptable contraception methods include at least one of the following: intrauterine (intrauterine device) or hormonal (oral, injection, patch, implant, ring) for at least 3 months, barrier with spermicide (condom, diaphragm), or abstinence.
7. Have pre-existing corneal astigmatism not exceeding 1.25 D in both eyes as determined by keratometry
8. Dilated pupil size 5.5 mm or greater to allow visualization of the IOL orientation marks post-operatively in both eyes

Eligible subjects must not meet any of the following exclusion criteria. Subjects may not participate if either eye meets any of the ocular exclusion criteria:

1. Previous intraocular, corneal, or retinal detachment surgery, including corneal transplant, LASIK / LASEK / PRK, SMILE, astigmatic keratotomy and limbal relaxing incisions in any eye
2. Diagnosed degenerative visual disorders (e.g. macular degeneration, retinal detachment, proliferative diabetic retinopathy, or other retinal disorders) that are predicted to cause future acuity losses to a level of 0.20 logMAR (20/30) or worse
3. Significant anterior segment pathology that might increase intraoperative risk or compromise IOL stability (e.g. pseudoexfoliation syndrome, any iris pathology)
4. Subjects with conditions associated with increased risk of zonular rupture (that may affect post-operative centration or tilt of IOL) in any eye
5. Potentially occludable angle or ciliary body tumor, or other pathology that might increase risk to subject safety, based on adequate diagnostics e.g. gonioscopic, anterior OCT observation
6. Subjects reasonably expected to require secondary ocular surgical intervention or laser treatment (other than YAG capsulotomy)
7. Subjects with clinically significant corneal pathology, potentially affecting corneal topography
8. Subjects with traumatic cataract in any eye
9. Currently participating in a drug or device clinical trial, or having participated in such a trial within 30 days prior to the pre-operative visit
10. Subjects with any other serious ocular pathology (e.g. severe dry eye, history of intraocular inflammation, history of retinal surgery or retinal laser procedure) or underlying systemic medical condition (e.g., uncontrolled diabetes) or circumstance that, based on the investigator's judgment, poses a concern for the subjects' safety or could confound the results of the study
11. Clinically significant, uncontrolled glaucoma with expected negative impact on IOL Rotational Stability and / or visual acuity outcomes in one or both eyes
12. Use of medications known to interfere with visual performance, pupil dilation, or iris structure within 30 days of the pre-operative visit, at the discretion of the investigator
13. Pregnant or nursing females
14. Pre-operative corneal astigmatism above 1.25D as determined by keratometry
15. Irregular astigmatism in any eye

    Additional Exclusion Criteria at the Time of Surgery:

    Subjects who do not meet exclusion criteria described in section 6.2 and are enrolled in the study may present findings during surgery that preclude inclusion of performance data in the investigation and thus need to be excluded from data collection post operatively. The following general exclusion criteria shall be considered during surgery for either eye:
16. zonular instability;
17. need for iris manipulation;
18. capsular fibrosis or other opacity;
19. inability to fixate IOL in desired position

If the IOL has touched the eye, it should be noted if the reason for exclusion is related to the IOL itself and/or any (e.g. IOL or insertion device defect causing capsular damage, malfunction of insertion device).

If the IOL has touched the eye, the subject should be followed, for safety, until completion of the investigation.

Min Age: 22 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 22 years or older who are scheduled for bilateral cataract surgery as part of routine clinical care and are in accordance with the study's inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoints - IOL axis misalignment | 120 to 150 days post-operatively (Visit 4)
  Percentage of RayOne Model RAO800S IOLs with IOL axis misalignment at Visit 4 (as determined by photographic method using baseline image at day of surgery) less than
  * 10 degrees in 90% of the cases as described in ISO 11979-7:2024.
  * 20 degrees in 95% of the cases as described in ISO 11979-7:2024.

SECONDARY OUTCOMES:
Secondary Effectiveness Endpoints - Stability of IOL axis orientation | 120 to 150 days post-operatively (Visit 4)
  Stability of IOL axis orientation, expressed as percentage of IOLs that rotate ≤ 5 degrees postoperatively between 30 to 60 days (Visit 3) and 120 to 150 days (Visit 4) as described in the ANSI Z80.30-2018. This criterium is passed if 90% of the IOLs in the treated eyes rotate ≤ 5 degrees between the mentioned visits.
Secondary Safety Endpoints - Rate of CDVA 0.30 logMAR | 120 to 150 days post-operatively (Visit 4)
  Rate of CDVA 0.30 logMAR or better at 120 to 150 days post-operatively (Visit 4) shall not exceed the ISO SPE threshold rates as described in ISO 11979-7:2024 (Table E.3)